CLINICAL TRIAL: NCT06608602
Title: The Pulmonary Effects of Tidal Volume Adjustment According to Forced Vital Capacity Versus Predicted Body Weight in Thoracic Surgery Patients
Brief Title: Tidal Volume Adjustment According to Forced Vital Capacity Versus Predicted Body Weight in Thoracic Surgery Patients
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, mediha turktan, dr, Cukurova University
Other Study IDs: TV01
Record Dates: First submitted 2024-09-11; First posted 2024-09-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-01

CONDITIONS: Thoracic Surgery; Tidal Volume; Forced Vital Capacity; Predicted Body Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group I and Group II: Group I= tidal volume 7 ml/predicted body weight Group II= tidal volume FVC/8 ml
  Interventions: Other: tidal volume adjustment during surgery

INTERVENTIONS:
Other: tidal volume adjustment during surgery — tidal volume adjustment during surgery according to body weight or FVC

SUMMARY:
The goal of this observational study is to learn about the intraoperative and postoperative pulmonary effects of tidal volume adjustment according to force vital capacity in thoracic surgery patients. The main question it aims to answer is:

Is there any positive effect of tidal volume adjustment according to force vital capacity on intraoperative and postoperative lung function in thoracic surgery patients?

Participants already taking tidal volume adjustment according to force vital capacity or predicted body weight during toracic surgery. As part of the medical care of thoracic surgery patients, intraoperative hemodynamic variables, lung dynamics and blood gas values and postoperative pulmonary complications will be monitored.

DETAILED DESCRIPTION:
Patients over 18 years of age and American Society of Anesthesiologists (ASA) physical status I-III who scheduled for elective thoracic surgery under general anesthesia will be included. Exclusion criteria: age > 18 years old, ASA I-III; III, pregnancy, presence of large bullae and/or pneumothorax, previous lung resection surgery, intensive care unit (ICU) admission in the preoperative period, predictive postoperative ICU admission, pneumonectomy surgery, and missing data.

In the operating room, all patients will be monitored with electrocardiogram, pulse oximeter, non-invasive arterial blood pressure. Anesthesia management, intraoperative and postoperative fluid management, postoperative analgesia regimens were will be standard procedures at the clinic for all patients.

During two-lung ventilation (TLV), mechanical ventilation will be set for a tidal volume (TV) of 7 ml/predicted body weight (PBW) for Group I, FVC/8 ml for Group II. Other settings will be similar between two groups; respiratory rate of 10-14 breaths/min, inspiratory time (Ti) of 33% without inspiratory pause.

Demographic data, functional status, ARISCAT score, hemodynamic values, respiratory measurements (peripheral oxygen saturation: SpO2, Ppeak, Pplato, TV, lung compliances, FiO2, end-tidal carbon dioxide: EtCO2), blood gas analysis (PaO2, PaCO2), and PaO2/ FiO2 rate will be recorded after intubation on TLV (T1), after lateral position on TLV (T2), after 30 min onset OLV (T3), the end of OLV on TLV (T4), and before extubation on TLV (T5).

Duration of anesthesia, duration of OLV, urine output, estimated blood loss, fluid therapy (ml, crystalloid and colloid), the need for blood product (ml), intraoperative complications, and the need for inotrope or vasopressor agent will also recorded during surgery.

The patients will be visited during postoperative five days (day 1: postoperative first day) and respiratory complications (pneumonia, pneumothorax, additional oxygen therapy, respiratory failure, acute respiratory distress syndrome, unplanned invasive or noninvasive mechanical ventilation, prolonged air leak, pleural effusion, atelectasis, cardiopulmonary edema) will be evaluated and recorded daily.

Length of hospital stay and in-hospital mortality will be also recorded. Hospitalization or intensive care unit admission within 30 days after surgery and mortality at 28 days will be assessed by calling the patients and their relatives by phone.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled for elective thoracic surgery under general anesthesia

Exclusion Criteria:

* Age over 18 years old,
* ASA > III,
* Pregnancy,
* Presence of large bullae and/or pneumothorax,
* Previous lung resection surgery,
* Intensive care unit (ICU) admission in the preoperative period,
* Predictive postoperative ICU admission,
* Pneumonectomy surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for elective thoracic surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
intraoperative oxygenation (PaO2/FiO2 ratio) | 5 time during surgery (T1:after intubation on TLV, T2: after lateral position on TLV, T3: after 30 min onset OLV, T4: the end of OLV on TLV, T5: before extubation on TLV
  The ratio of partial pressure of oxygen in arterial blood (PaO2) to the fraction of inspiratory oxygen concentration (FiO2) is an indicator of pulmonary shunt fraction.
lung compliance (mL/cmH2O) | 5 time during surgery (T1:after intubation on TLV, T2: after lateral position on TLV, T3: after 30 min onset OLV, T4: the end of OLV on TLV, T5: before extubation on TLV
  static and dynamic compliance

SECONDARY OUTCOMES:
postoperative pulmonary complications | Through postoperative 5 days
  Postoperative pulmonary complications were defined pneumonia, pneumothorax, additional oxygen therapy, respiratory failure, acute respiratory distress syndrome, unplanned invasive or noninvasive mechanical ventilation, prolonged air leak, pleural effusion, atelectasis, and cardiopulmonary edema.
Length of hospital stay (day) | Through postoperative period, an avarage of 5 days
  from the day of surgery until the day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: mediha Turktan, MD, Principal Investigator — Cukurova University
Locations (2):
- Turkey (Türkiye) (2):
  - Cukurova University Faculty of Medicine Anesthesiology Department, Adana, Adana
  - Cukurova University Faculty of Medicine Anesthesiology Department, Adana

IPD SHARING:
Plan to Share IPD: Undecided